CLINICAL TRIAL: NCT06771921
Title: First-in-Human, Open-Label, Dose-Escalation Trial With Expansion Cohorts to Evaluate Safety and Preliminary Efficacy of GEN1078 in Subjects With Malignant Solid Tumors
Brief Title: A First-in-Human Trial of Safety and Efficacy of GEN1078 in Participants With Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The sponsor has made the decision to terminate further development of GEN1078 based on emerging safety observations and overall benefit-risk assessment of 1078
Sponsor: Genmab (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GCT1078-01; 2024-515752-21-00 (EU CTIS Number)
Record Dates: First submitted 2025-01-08; First posted 2025-01-13 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Malignant Solid Tumor

STUDY DESIGN:
Intervention Model Description: No randomization will be performed in the Dose-escalation part. In Dose-expansion part, if two expansion doses are identified, participants will be randomized to either Expansion Dose 1 or Expansion Dose 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose-Escalation (Experimental): GEN1078 will be administered as monotherapy until one of the treatment discontinuation criteria has been met.
  Interventions: Drug: GEN1078
- Dose Expansion (Experimental): GEN1078 will be administered as monotherapy until one of the treatment discontinuation criteria has been met.
  Interventions: Drug: GEN1078

INTERVENTIONS:
Drug: GEN1078 — Specified dose on specified days.

SUMMARY:
The purpose of this trial is to measure the following in participants with solid cancers who receive GEN1078.

* The side effects seen with GEN1078
* What the body does with GEN1078 once it is administered
* What GEN1078 does to the body once it is administered
* How well GEN1078 works against advanced solid tumors

Trial details include:

* The estimated trial duration is 8 months for an individual participant (the trial duration may vary for each participant).
* The treatment duration will be an estimated 3-month treatment period (the duration of treatment may vary for each participant).
* The visit frequency will be daily or visits every few days for the first few months.

All participants will receive active drug; no one will be given placebo.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have at least 1 measurable lesion per RECIST v1.1 assessed by the investigator.
* Must have an Eastern Cooperative Oncology Group performance status (ECOG PS) score of 0 to 1.

Dose Escalation Only

* Participant must have histologically or cytologically confirmed solid tumor(s) for which there is no further available standard therapy likely to confer clinical benefit (or participant is not a candidate or has previously refused such earlier available therapy), and for whom, in the opinion of the investigator, experimental therapy with GEN1078 may be beneficial.
* Must have either recurrence after, or progression on available relevant standard of care (SoC) anticancer therapies; or are deemed intolerant to or ineligible for, standard curative therapy in the recurrent setting.

Expansion Only

* Participant must have advanced (unresectable) or metastatic, histologically confirmed diagnosis of selected solid cancers.

Key Exclusion Criteria:

* Has significant cardiovascular impairment within 6 months prior to the first dose of trial drug, including presence of unstable angina, myocardial infarction, congestive heart failure (New York Heart Association [NYHA] class III and IV), or clinically significant cardiac arrhythmia (other than stable atrial fibrillation) requiring anti-arrhythmia therapy.
* Known unstable central nervous system (CNS) metastases or any active or history of carcinomatous meningitis.
* Has been exposed to any of the following prior therapies within the specified timeframes:

  * Prior therapy with a compound targeting the same targets as GEN1078 or any cell-based therapies.
  * Radiotherapy within 14 days prior to C1D1. Palliative radiotherapy of bone metastases up to 7 days prior to C1D1 will be allowed.
  * Treatment with any investigational or non-investigational anticancer agent (including investigational vaccines) or used an invasive investigational medical device within 28 days or 5 half-lives of the drug, whichever is shorter, prior to the first dose of GEN1078.
  * Chemotherapy within 2 weeks prior to the first dose of GEN1078.
  * Prophylaxis with live, attenuated vaccines within 28 days prior to first dose of GEN1078; or prophylaxis with the first and/or subsequent injection(s) of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) nucleic acid vaccine within 14 days prior to first dose of GEN1078.
  * Chronic systemic immunosuppressive treatment, including corticosteroids, ie, prednisone >10 milligrams (mg) daily (or equivalent) or a cumulative dose >140 mg prednisone within 14 days (or equivalent) before the first dose of GEN1078. Replacement therapy (eg, physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is permitted.
  * Has received granulocyte colony-stimulating factor (G-CSF) or granulocyte/macrophage colony stimulating factor support within 2 weeks prior to the first dose GEN1078 or being chronically transfusion dependent.
  * Has received other T-cell activating surface marker. Note: Prior treatment with anti-T-cell Ig and ITIM domain (aTIGIT), anti-programmed cell death protein 1 (aPD1), anti-programmed death-ligand 1 (aPDL1), anti-lymphocyte activation gene 3 protein (aLAG3), anti-cytotoxic T-lymphocyte-associated protein 4 (aCTLA-4) is allowed.
  * The initiation of growth factors and bisphosphonates is not allowed during the first 4 weeks of GEN1078 administration, unless agreed upon by the investigator and sponsor medical monitor. However, the use of receptor activator of nuclear factor kappa-Β ligand (RANK-L) inhibitors and bisphosphonates (if on stable dose for at least 4 weeks) is permitted while participating in this trial.

NOTE: Other protocol-defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2025-01-29 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
Dose Escalation: Number of Participants With Dose-limiting Toxicities (DLTs) | Up to 21 days
  Toxicities will be graded for severity according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) criteria version 5.0, except for cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS) which will be evaluated according to the American Society for Transplantation and Cellular Therapy (ASTCT) criteria.
Dose Escalation: Number of Participants With Adverse Events (AEs) | From first dose until the end of the safety follow-up period (30 days after the last dose)
Dose Expansion: Confirmed Objective Response Rate (ORR) | Up to approximately 5 years
  Confirmed ORR is defined as the percentage of participants with confirmed best overall response (BOR) of complete response (CR) or partial response (PR) based on response evaluation criteria in solid tumors (RECIST) v1.1 as assessed by the investigator.

SECONDARY OUTCOMES:
Dose-Escalation and Expansion: Clearance (CL) of GEN1078 | Predose and postdose at multiple timepoints up to end of treatment (approximately 3 months)
Dose-Escalation and Expansion: Volume of Distribution (Vd) of GEN1078 | Predose and postdose at multiple timepoints up to end of treatment (approximately 3 months)
Dose-Escalation and Expansion: Area Under the Concentration-Time Curve from Time Zero to Last Quantifiable Concentration (AUC0-last) of GEN1078 | Predose and postdose at multiple timepoints up to end of treatment (approximately 3 months)
Dose-Escalation and Expansion: Area Under the Concentration-Time Curve from Time Zero to Infinity (AUC0-∞) of GEN1078 | Predose and postdose at multiple timepoints up to end of treatment (approximately 3 months)
Dose-Escalation and Expansion: Maximum Observed Plasma Concentration (Cmax) of GEN1078 | Predose and postdose at multiple timepoints up to end of treatment (approximately 3 months)
Dose-Escalation and Expansion: Time to Reach Cmax (Tmax) for GEN1078 | Predose and postdose at multiple timepoints up to end of treatment (approximately 3 months)
Dose-Escalation and Expansion: Predose Concentration for GEN1078 | Predose up to end of treatment (approximately 3 months)
Dose-Escalation and Expansion: Terminal Half-life (t½) of GEN1078 | Predose and postdose at multiple timepoints up to end of treatment (approximately 3 months)
Dose-Escalation and Expansion: Number of Participants with Anti-drug Antibodies (ADAs) | Up to approximately 5 years
Dose Escalation: Confirmed ORR | Up to approximately 5 years
  Confirmed ORR is defined as the percentage of participants with confirmed BOR of CR or PR based on RECIST v1.1 as assessed by the investigator.
Dose-Escalation and Expansion: Duration of Response (DOR) | Up to approximately 5 years
  DOR is defined as the time from first documentation of response (CR or PR) to the date of the first documented progression or death whichever occurs earlier based on RECIST v1.1 as assessed by the investigator.
Dose-Escalation and Expansion: Disease Control Rate (DCR) | Up to approximately 5 years
  The DCR is defined as the percentage of participants with confirmed BOR of CR, PR, or Stable Disease (SD) according to RECIST v1.1 as assessed by investigator.
Dose-Escalation and Expansion: Time to Response (TTR) | Up to approximately 5 years
  TTR based on investigator assessment is defined as the time from Cycle 1, Day 1 (C1D1) to first documentation of objective response (CR or PR) in participants achieving PR or CR according to RECIST v1.1 as assessed by investigator.
Dose Expansion: Number of Participants With AEs | From first dose until the end of the safety follow-up period (30 or 60 days after the last dose)

CONTACTS AND LOCATIONS:
Overall Officials: Study Official, Study Director — Genmab
Locations (6):
- Righshospitalet (Copenhagen University Hospital), Copenhagen, Denmark
- Spain (5):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Centro Integral Oncologico Clara Campal, Madrid
  - Hospital Universitary Fundacion Jimenez Diaz, Madrid
  - NEXT Oncology Madrid, Madrid
  - Clinica Universidad de Navarra, Pamplona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results Summary in Plain Language — https://euclinicaltrials.eu/search-for-clinical-trials/?lang=en&EUCT=2024-515752-21-00